CLINICAL TRIAL: NCT00667004
Title: Efficacy Study of Ecabet Ophthalmic Solution in Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-S&E-1107071-P
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ecabet ophthalmic solution
  Interventions: Drug: ecabet ophthalmic solution
- 2 (Placebo Comparator): Placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ecabet ophthalmic solution — sterile ophthalmic solution
  Arms: 1
Drug: placebo — sterile ophthalmic solution
  Arms: 2

SUMMARY:
Efficacy study of ecabet ophthalmic solution in dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dry eye disease

Exclusion Criteria:

* Dry eye disease secondary to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2008-03-22 (Actual); Primary Completion 2008-09-12 (Actual); Study Completion 2008-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ecabet Ophthalmic Solution: ecabet ophthalmic solution
  ecabet ophthalmic solution: sterile ophthalmic solution
- Vehicle: Placebo comparator
  placebo: sterile ophthalmic solution
Period: Overall Study
Arm/Group | Ecabet Ophthalmic Solution | Vehicle
Started | 95 | 88
Completed | 93 | 85
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecabet Ophthalmic Solution | Vehicle | Total
Number analyzed (Participants) | 95 | 88 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (13.2) | 56.0 (15.2) | 56.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 63 | 139
  Male | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Lacrimation Assessed by Schirmer's Test
Description: The Schirmer's test is used determine if tear glands produce enough tears to keep eyes adequately moist. Calibrated strips of a non-toxic filter paper are used. One free end is placed within the lower eyelid. At the conclusion of the test, the paper strip is removed from the lower eyelid and the amount of wetting of the paper strip is measured.
Time Frame: 43 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ecabet Ophthalmic Solution | Vehicle
Number analyzed (Participants) | 95 | 88
mm
  Anesthetized | 3.02 (4.70) | 2.15 (4.40)
  Unanesthetized | 2.35 (5.53) | 1.35 (5.38)

ADVERSE EVENTS:
Time Frame: 43 days
Arm/Group | Ecabet Ophthalmic Solution | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/95 | 0/88
Other Adverse Events (participants affected / at risk) | 0/95 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ecabet Ophthalmic Solution (N=95) | Vehicle (N=88)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.